CLINICAL TRIAL: NCT00478218
Title: A Phase II Trial of Revlimid, Cyclophosphamide, and Dexamethasone in Patients With > Newly Diagnosed Active Multiple Myeloma
Brief Title: Lenalidomide, Cyclophosphamide, and Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546657; P30CA015083 (NIH); MC058E (Other: Mayo Clinic Cancer Center); 06-002786 (Other: Mayo Clinic IRB); RV-MM-PI-0116 (Other: Celgene Protocol)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2011-07-27 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide/Cyclophosphamide/Dexamethasone (Experimental)
  Interventions: Drug: cyclophosphamide; Drug: dexamethasone; Drug: lenalidomide

INTERVENTIONS:
Drug: cyclophosphamide — 300 mg/m2 administrated by PO (with food)on Days 1, 8, 15 (up to 12 cycles) OR 300 mg administrated by PO (with food)on Days 1, 8, 15 (up to 12 cycles)
  Other Names: Cytoxan, CTX, Neosar®
Drug: dexamethasone — 40 mg administrated by PO (with food)on Days 1, 8, 15 & 22
  Other Names: Decadron
Drug: lenalidomide — 25 mg administrated by PO (with food)on Days 1-21
  Other Names: Revlimid®

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with cyclophosphamide and dexamethasone may kill more cancer cells.> PURPOSE: This phase II trial is studying how well giving lenalidomide together with cyclophosphamide and dexamethasone works in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the response rate in patients with newly diagnosed active multiple myeloma treated with lenalidomide, cyclophosphamide, and dexamethasone.

Secondary

* Assess the toxicity of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen. OUTLINE: Patients receive oral lenalidomide on days 1-21, oral cyclophosphamide on days 1, 8, and 15, and oral dexamethasone on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4-12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Newly diagnosed disease
  * Symptomatic disease
* Measurable or evaluable disease, defined by ≥ 1 of the following criteria:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * Monoclonal protein > 200 mg by 24-hour urine electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (evaluable disease)
  * Measurable soft tissue plasmacytoma not previously irradiated
* No monoclonal gammopathy of undetermined significance or smoldering myeloma

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 (ECOG PS 3 allowed if secondary to pain)
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Creatinine ≤ 2.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception (1 highly effective and 1 additional method) for 1 month before, during, and for 4 weeks after completion of study therapy
* No uncontrolled infection
* No other active malignancy
* No other malignancies within the past 5 years except for currently treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* No NYHA class III-IV congestive heart failure
* No untreated active deep vein thrombosis

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior radiotherapy for solitary plasmacytoma
* Prior clarithromycin, therapeutic dehydroepiandrosterone (DHEA), anakinra, pamidronate disodium, or zoledronic acid allowed
* No prior cytotoxic chemotherapy
* No prior corticosteroids (except for treatment of a nonmalignant disorder)
* Concurrent corticosteroids (prednisone ≤ 20 mg/per day) allowed
* No concurrent radiotherapy except palliative radiotherapy for a single painful bone lesion or fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Study Chair — Mayo Clinic; Craig B. Reeder, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic Cancer Center, Rochester, Minnesota

REFERENCES:
- [Result] Kumar SK, Lacy MQ, Hayman SR, Stewart K, Buadi FK, Allred J, Laumann K, Greipp PR, Lust JA, Gertz MA, Zeldenrust SR, Bergsagel PL, Reeder CB, Witzig TE, Fonseca R, Russell SJ, Mikhael JR, Dingli D, Rajkumar SV, Dispenzieri A. Lenalidomide, cyclophosphamide and dexamethasone (CRd) for newly diagnosed multiple myeloma: results from a phase 2 trial. Am J Hematol. 2011 Aug;86(8):640-5. doi: 10.1002/ajh.22053. Epub 2011 May 31. PMID 21630308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-three (53) participants were recruited between July 2006 and August 2008 at Mayo Clinic.
Groups:
- LCD (Cyclophosphamide 300 mg/m^2): Lenalidomide 25 mg PI days 1-21 Cyclophosphamide 300 mg/m^2 PO days 1, 8, 15 Dexamethasone 40 mg PI days 1, 8, 15, 22
- LCD (Cyclophosphamide 300 mg): Lenalidomide 25 mg PI days 1-21 Cyclophosphamide 300 mg PO days 1, 8, 15 Dexamethasone 40 mg PI days 1, 8, 15, 22
Period: Overall Study
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg)
Started | 34 | 19
Completed | 34 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg) | Total
Number analyzed (Participants) | 34 | 19 | 53
Age Continuous [Median (Full Range); unit: years] | 63.5 [44 to 79] | 65 [37 to 82] | 64 [37 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 17 | 10 | 27
Region of Enrollment [Number; unit: participants]
  United States | 34 | 19 | 53
Durie Salmon Stage [Number; unit: paricipants]
  Stage IA - Low Cell Mass | 3 | 1 | 4
  Stage IIA - Intermediate Cell Mass | 7 | 11 | 18
  Stage IIIA/B - High Cell Mass | 24 | 7 | 31
Parameter of Hematologic Response - Serum M-spike >= 1 g/dL [Number; unit: participants]
  Yes | 25 | 14 | 39
  No | 9 | 5 | 14
Parameter of Hematologic Response - Serum Immunoglobulin Free Light Chain >= 10 mg/dL [Number; unit: participants]
  Yes | 21 | 14 | 35
  No | 13 | 5 | 18
Parameter of Hematologic Response - Urine M-Spike >= 200 mg/24 hours [Number; unit: participants]
  Yes | 11 | 5 | 16
  No | 23 | 14 | 37
Parameter of Hematologic Response - Bone Marrow Plasma Cells > 30% [Number; unit: participants]
  Yes | 17 | 14 | 31
  No | 17 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Confirmed Response (CR), Very Good Partial Response (VGPR) or Partial Response (PR) During Treatment
Description: Response that was confirmed on 2 consecutive evaluations during treatment
  * Complete Response(CR): Complete disappearance of M-protein from serum & urine on immunofixation, normalization of Free Light Chain (FLC) ratio & <5% plasma cells in bone marrow (BM)
  * Very Good Partial Response(VGPR): >=90% reduction in serum M-component; Urine M-Component <100 mg per 24 hours; <=5% plasma cells in BM
  * Partial Response PR): >= 50% reduction in serum M-Component and/or Urine M-Component >= 90% reduction or <200 mg per 24 hours; or >= 50% decrease in difference between involved and uninvolved FLC levels
Time Frame: Duration of Treatment (up to 5 years)
Measure: Number; unit: participants
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg)
Number analyzed (Participants) | 34 | 19
participants | 28 | 16

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from registration to death of any cause. Participants were followed for a maximum of 5 years from randomization. The median OS with 95%CI was estimated using the Kaplan Meier method.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg)
Number analyzed (Participants) | 34 | 19
months | NA [NA to NA] — Median OS for group 1 has not been attained. | NA [NA to NA] — Median OS for group 2 has not been attained.

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from registration to progression or death due to any cause. The median PFS with 95%CI was estimated using the Kaplan Meier method.> Progression was defined as any one or more of the following:> An increase of 25% from lowest confirmed response in:>
  * Serum M-component (absolute increase >= 0.5g/dl)>
  * Urine M-component (absolute increase >= 200mg/24hour>
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl>
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg)
Number analyzed (Participants) | 34 | 19
months | 27 [14 to 32.6] | NA [NA to NA] — The median PFS for group 2 has not been attained

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was calculated from the documentation (date) of first response (CR, VGPR, or PR) until the date of progression or last follow-up in the subset of patients who responded. The median DOR with 95%CI was estimated using the Kaplan Meier method.
Time Frame: up to 5 years
Population: Participants who achieved a partial response(PR) or better were evaluable for this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg)
Number analyzed (Participants) | 26 | 16
months | 26.1 [17.5 to 31.7] | NA [NA to NA] — Median DOR for group 2 has not been attained.

ADVERSE EVENTS:
Arm/Group | LCD (Cyclophosphamide 300 mg/m^2) | LCD (Cyclophosphamide 300 mg)
Serious Adverse Events (participants affected / at risk) | 13/34 | 2/19
Other Adverse Events (participants affected / at risk) | 34/34 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCD (Cyclophosphamide 300 mg/m^2) (N=34) | LCD (Cyclophosphamide 300 mg) (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Lung (pneumonia) infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin (cellulites) infection (Infections and infestations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 2 (2) | 0 (0)
Neutropenia (Investigations) | 5 (5) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ischemia-Cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCD (Cyclophosphamide 300 mg/m^2) (N=34) | LCD (Cyclophosphamide 300 mg) (N=19)
Anemia (Blood and lymphatic system disorders) | 14 (50) | 10 (37)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Diarrhea-No Colostom (Gastrointestinal disorders) | 7 (17) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Oral cavity Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain-Abdominal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Edema: Limb (General disorders) | 3 (5) | 1 (1)
Fatigue (General disorders) | 31 (239) | 18 (174)
Fever-No ANC (General disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Skin (cellulites) infection (Infections and infestations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 21 (96) | 14 (67)
Lymphopenia (Investigations) | 2 (24) | 4 (24)
Neutropenia (Investigations) | 31 (288) | 16 (163)
Platelet count decreased (Investigations) | 19 (70) | 12 (86)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (8) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 0 (0)
Extremity-lower weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Extremity-upper weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (61) | 14 (108)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope Vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (3)
Agitation (Psychiatric disorders) | 4 (8) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (8) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3) | 0 (0)
Depression (Psychiatric disorders) | 4 (5) | 2 (2)
Euphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (12) | 4 (6)
Cystitis (Renal and urinary disorders) | 6 (8) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Impotence (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (8)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes